CLINICAL TRIAL: NCT01159977
Title: Trial Evaluating the Effect of Facilitated Small Group Sessions on Physician Well-Being, Job Satisfaction, and Professionalism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Colin West, Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-008232
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Physician Well-being; Physician Job Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Facilitated small group (Experimental): Facilitated small groups.
  Interventions: Behavioral: Facilitated small groups
- Unstructured protected time (Active Comparator): Same time provided as for facilitated small groups, but without structure.
  Interventions: Behavioral: Unstructured time.
- Usual practice (Placebo Comparator): No protected time.
  Interventions: Behavioral: Usual practice

INTERVENTIONS:
Behavioral: Facilitated small groups — 1 hour sessions every 2 weeks for small groups of 9 participants, 19 sessions over 9 months.
  Arms: Facilitated small group
Behavioral: Unstructured time. — 1 protected hour every 2 weeks for 9 months, without small group structure.
  Arms: Unstructured protected time
Behavioral: Usual practice — No protected time provided.
  Arms: Usual practice

SUMMARY:
The study purpose is to evaluate the effect of a small group discussion based intervention on physician well-being, job satisfaction, and professionalism. Participants will be put in one of 3 groups by chance (as in the flip of a coin). A computerized selection process will be used to assign participants to the study groups. There is a 1 in 3 chance of being assigned at random to either of the 3 groups.

The first study group will meet once every two weeks for 9 months (from September 2010 through June 2011) from 12:30 pm until 2:00 pm. These meetings will be small group discussion sessions with groups of no more than 15 participants. Lunch will be provided for the first 30 minutes, and group discussion during the next 1 hour will be guided by the session facilitator around such topics as work-life balance, meaning in work, medical mistakes, spirituality, and unmet patient needs. However, the discussions will be open forums, and the groups themselves will help decide on topics relevant to the group. The 1 hour of protected non-clinical time every other week required for this group will be funded by the study.

The second study group will also have 1 hour of protected non-clinical time provided every other week for the same 9 months. This study group will not participate in small group discussions, but may use the protected time for professional tasks as they wish.

Participants in the third study group will continue with their current work practices, but will be provided with protected time to complete study surveys. If group sizes are too small after recruitment to allow a complete study of all three groups, the third study group will be removed and participants will be randomly assigned to one of the first two study groups only.

Participants in all groups will be asked to complete a quarterly survey on well-being, job satisfaction, and professionalism. Follow-up surveys will also be administered 3 months and 1 year after the conclusion of the small group sessions. Each survey is expected to take approximately 20-30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Senior Associate Consultant or Consultant in the Mayo Clinic Department of Medicine.

Exclusion Criteria:

* No clinical effort.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Physician burnout | September 2010 - June 2012
  Burnout measured by the Maslach Burnout Inventory.

SECONDARY OUTCOMES:
Physician job satisfaction | September 2010 - June 2012
  Job satisfaction measured by validated scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493